CLINICAL TRIAL: NCT02774018
Title: Life Satisfaction and Psychopathology in Institutionalized Elderly People: The Results of an Adapted Mindfulness-Based Stress Reduction Program
Brief Title: Life Satisfaction and Psychopathology in Institutionalized Elderly People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Irmandade da Misericórdia de Albergaria-a-Velha (Other)
Responsible Party: Principal Investigator, Daniel Seabra, Investigator, Irmandade da Misericórdia de Albergaria-a-Velha
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 01_PSI_MINDFULNESS
Record Dates: First submitted 2016-04-18; First posted 2016-05-16 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Anxiety Depression (Mild or Not Persistent)
Keywords: Mindfulness; Elderly; Psychopathology
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Mindfulness-Based Stress Reduction

ARMS (1):
- 12 institutionalized elderly people (Experimental): Mindfulness-Based Stress Reduction program.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction (MBSR) program

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction (MBSR) program

SUMMARY:
The present study attempted to test the benefits of a Mindfulness-Based Stress Reduction (MBSR) program in Portuguese institutionalized elderly people, as a way to improve life satisfaction and reduce psychopathology. The sample included 12 institutionalized elderly people, with ages between 65 and 91 (M = 82.58 years; SD = 7.87), that filled several selfreport questionnaires and were assessed with Mini Mental State Examination. Participants attended to an adapted Mindfulness-Based Stress Reduction program (KabatZinn,1994), with 48 sessions (16 weeks) and Participants were evaluated before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* literacy
* age above 65 years

Exclusion Criteria:

* presence of cognitive or sensorial
* impairment

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in depression levels assessed with the GDS | Pre-test and Post-test (4 months later)
  GDS; Geriatric Depression Scale; Greenberg et al., 2005
Change in anxiety levels assessed with the DASS-21 | Pre-test and Post-test (4 months later)
  DASS-21; Depression Anxiety Stress Scale; Lovibond e Lovibond, 1995
Change in experiential avoidance levels assessed with the AAQ-II | Pre-test and Post-test (4 months later)
  AAQ-II; Acceptance and Action Questionnaire; Bond, Hayes, Baer, Carpenter, Guenole, Orcutt, Waltz e Zettle, 2011
Change in subjective pain levels assessed with the Faces Scale | Pre-test and Post-test (4 months later)
  Faces Scale; Wong et al., 2001
Change in life satisfaction levels assessed with the SWLS | Pre-test and Post-test (4 months later)
  SWLS; Satisfaction with Life Scale; Diener et al., 1985